CLINICAL TRIAL: NCT04469023
Title: Late Phase II Study of TS-142 in Patients with Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TS142-203
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2021-12

CONDITIONS: Patients with Insomnia
MeSH Terms: interventions — TS-142

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TS-142 2.5 mg (Experimental): Period in which participants received multiple-dose of 2.5 mg TS-142 prior to bedtime
  Interventions: Drug: TS-142
- TS-142 5 mg (Experimental): Period in which participants received multiple-dose of 5 mg TS-142 prior to bedtime
  Interventions: Drug: TS-142
- TS-142 10 mg (Experimental): Period in which participants received multiple-dose of 10 mg TS-142 prior to bedtime
  Interventions: Drug: TS-142
- Placebo (Experimental): Period in which participants received single placebo prior to bedtime
  Interventions: Drug: TS-142

INTERVENTIONS:
Drug: TS-142 — Participants received multiple-dose of 2.5, 5, 10 mg of TS-142 or placebo (oral tablet)

SUMMARY:
This is a randomized, double-blind, multi-center, placebo-controlled, parallel-group exploratory study in patients with insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male and female age 20 years or older at the time of informed consent
* Outpatients
* Patients who meet the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria for insomnia disorder
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Patients who meet the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria excepting insomnia disorder preceding visit 1
* Patients who meet the DSM-5 criteria for Restless legs syndrome at visit 1
* Patients with comorbid psychiatric disorder(s), including depression, schizophrenia, anxiety
* Other protocol defined exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
LS mean difference from placebo; Change between baseline and end of the study of sSL | Baseline and Week 2
  sSL is defined as the duration of time that it took to fall asleep as recorded in a sleep diary

SECONDARY OUTCOMES:
LS mean difference from placebo; Change between baseline and end of the study of sTST | Baseline and Week 2
  sTST is defined as the total amount of time spent asleep before getting-out from his/her bed for the day as recorded in a sleep diary
LS mean difference from placebo; Change between baseline and end of the study of sWASO | Baseline and Week 2
  sWASO is defined as the total amount of time spent awake after falling asleep and before getting-out from bed for the day as recorded in a sleep diary.

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No